CLINICAL TRIAL: NCT00532025
Title: A Phase II Study to Investigate the Efficacy and Safety of Sorafenib as Adjuvant Treatment Following Resection of Non-small Cell Lung Carcinoma (NSCLC) in Patients Not Eligible for Cisplatin-based Adjuvant Chemotherapy
Brief Title: Sorafenib in Resected Non-small Cell Lung Carcinoma
Acronym: SIRN
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Prof. Martin Schuler, University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIRN-TOM1 KKS 2006-010
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Last update posted 2009-07-28 (Estimated); Status verified 2009-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Sorafenib; NSCLC; Adjuvant Treatment; resected Non-Small Cell Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Sorafenib treatment
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — Sorafenib will be administered as oral formulation (200 mg tablets) at a dose of 400 mg twice daily starting 28 to 42 days after surgery or surgery plus adjuvant radiotherapy. The dose may be adjusted based on individual toxicities following a predetermined dose reduction schedule. Sorafenib therapy will be continued for 48 months, or until disease progression, patient refusal or intolerable toxicity, whichever comes first. Patients in remission after 48 months will be offered continued Sorafenib treatment in a roll-over study.
  Other Names: Nexavar

SUMMARY:
This is an open-label, single-armed, multicentric, phase II study of Sorafenib treatment following surgery for NSCLC.

The primary hypothesis is to increase the progression-free survival (PFS) of the experimental group in comparison to a historical control group. For sample size calculation a 2 year PFS of 50% was calculated for the historical control group, and a 2 year PFS of 67% was estimated for the intervention group. These estimates are based on the actual PFS and overall survival (OS) of a defined population of 120 NSCLC patients treated at a single institution with surgery alone or surgery followed by adjuvant radiotherapy, which compares favorably to published international results, and the improvement of PFS achieved by 4 cycles of cisplatin/vinorelbine-based cytotoxic chemotherapy in published randomized trials.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed diagnosis of NSCLC pathological stages I, II or III A
* Patients must have completely resected disease and may not be treated with prior chemotherapy. Patients must have fully recovered from surgery prior to initiation of study treatment.
* Adjuvant radiotherapy for stage III A disease is permitted given that the patient has recovered from all radiation-induced toxicities. In those patients, a complete restaging will be performed prior to enrolment into the trial.
* Patients with completely resected NSCLC stage II or III A, who for medical reasons are not eligible for adjuvant chemotherapy consisting of a standard regimen of 4 cycles cisplatin/vinorelbine
* Patients with completely resected NSCLC stage II or III A, who are not willing to undergo adjuvant chemotherapy with 4 cycles of cisplatin/ vinorelbine, are also eligible.
* Age ≥ 18 years
* ECOG performance status ≤ 2
* Normal organ and marrow function defined as:

Hematopoetic: absolute neutrophil count >1,500/mm3, platelet count > 100,000/mm3, hemoglobin > 9 g/dL INR < 1.5 ULN and PTT within normal limits Hepatic: total bilirubin < 1.5 x ULN, AST or ALT < 2.5 x ULN Renal: creatinine < 1.5 x ULN

* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment
* Women of childbearing potential and men must agree to use adequate birth contraception prior to study entry and for the duration of study participation. Women and men should use adequate birth control for at least 3 months after the last administration of Sorafenib.
* Written informed consent

Exclusion Criteria:

* Any other histology (e.g. SCLC, carcinoid tumors) or disease stages other than I to III A
* Patients who are eligible and willing to undergo a standard adjuvant chemotherapy regimen (4 cycles of cisplatin/vinorelbine)
* Any prior systemic anticancer therapy including chemotherapy, targeted agents, experimental therapy or biological therapy for NSCLC
* Cardiac disease: congestive heart failure > class II NYHA, patients must not have unstable angina pectoris or new onset of angina pectoris or myocardial infarction within the past 6 months, or cardiac ventricular arrhythmias requiring antiarrhythmic therapy
* Uncontrolled hypertension defined as systolic blood pressure > 150 mm Hg or diastolic pressure > 90 mm Hg, despite optimal therapy
* Known brain metastasis. Patients with symptoms should undergo CT scan/MRI of the brain to exclude brain metastasis
* Active clinically serious infections > NCI-CTCAE Grade 2
* Thrombotic or embolic events including transient ischemic attacks within the past 6 months
* Hemorrhage/bleeding event ≥ NCI-CTCAE Grade 3 within 4 weeks before first dose of study drug
* Serious non-healing wound, ulcer or bone fracture
* Evidence or history of bleeding diathesis or coagulopathy
* Therapeutic anticoagulation with Vitamin K antagonists such as warfarin, phenprocoumon, or with heparins or heparinoids. Low dose warfarin/phenprocoumon is permitted if INR is < 1.5. Low dose aspirin (300 mg/d) is permitted.
* Use of St John's Wort or rifampicin
* Major surgery, open biopsy or significant traumatic injury within 4 weeks before first dose of study drug
* Known or suspected allergy to Sorafenib or any agent given in the course of this trial
* Previous cancer that is distinct in primary site or histology from NSCLC except cervical cancer in situ, treated basal cell carcinoma, superficial bladder tumors or any cancer curatively treated ≥ 3 years prior to study entry.
* Substance abuse, medical or psychological condition that may interfere with the patient´s participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) clinical and radiological assessment of remission status (RECIST criteria) | 2 years

SECONDARY OUTCOMES:
Progression free survival | 3 and 4 years
Overall survival | 3 and 4 years
Assessment of safety and tolerability of Sorafenib when administered as adjuvant treatment following surgery for NSCLC | 2, 3 and 4 years
Assessment of biomarkers relevant to Sorafenib response and disease state, and their correlation to clinical outcome | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schuler, MD, Principal Investigator — Innere Klinik (Tumorforschung), Westdeutsches Tumorzentrum, Universitätsklinikum Essen, Hufelandstrasse 55, 45122 Essen
Locations (6):
- Germany (6):
  - SIRN investigational trial site, Essen
  - SIRN investigational trial site, Halle
  - SIRN investigational trial site, Löwenstein
  - SIRN investigational trial site Johannes Gutenberg Universität, Mainz
  - SIRN investigational trial site Katholisches Klinikum, Mainz
  - SIRN investigational trial site, Rotenburg (Wümme)